CLINICAL TRIAL: NCT00363532
Title: Functional MRI (fMRI) in Patients With Migraine Without Aura Provoked by
Brief Title: Functional MRI (fMRI) in CGRP Induced Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Mohammad Sohail Asghar, MD, Neurological Dep. University of Copenhagen, Denmark, Glostrup Hospital.
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KA-20060083
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Migraine Without Aura
Keywords: migraine with out aura
MeSH Terms: conditions — Migraine without Aura

INTERVENTIONS:
Drug: infusion of calcitonin gene related peptide (CGRP)

SUMMARY:
In patients known with migraine without aura a migraine headache or migraine like headache will be induced by infusion of calcitonin gene related peptide (CGRP). The patients will then be stimulated with noxious heat via a thermode placed at the forehead. At the same time the Blood-oxygenation-level-dependent (BOLD) response will be measured via functional magnetic resonance imaging (fMRI), to estimate the central-nervous pain response. The regions of interest (ROI) will be thalamic region and medulla oblongata.

Then the patients will be given pain relif in form of injection of sumatriptan and the effect of this will also be registered via measuring the BOLD response at the RIO's previously defined. A 3-Tesla MRI scanner will be used in this trail.

This study will give us key knowledge of the trigeminal pain pathway and the central processing i.e sensitization during a migraine attach.

ELIGIBILITY:
Inclusion Criteria:

* Patients know with migraine without aura.
* No less then 1 migraine attach pr month and no more then 6 attaches per month.
* Weight 50-100 kg.
* Women must be using secure birthcontrol.

Exclusion Criteria:

* Tension type headache more then 1 day/month.
* All other prim. og sec. headache types then migraine without aura.
* Daily use of medication other then birthcontrol pills.
* Pregnant and lactation women.
* Headache on the trail day or 5 days previous to the trail day.
* Contraindications to MRI-scans.
* Hypertension or hypotension.
* Known heart or lung condition.
* Mental illness or substance abuse.
* Other considerable conditions judged by the including doctor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Changes in BOLD response before and after CGRP infusion.
Changes in BOLD response before and after injection of sumatriptan.

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, MD,PH.d, Study Chair — Danish Headache Center
Locations (1):
- Danish Headache Center, Neurological Dep. Glostrup hospital, Glostrup Municipality, Denmark